CLINICAL TRIAL: NCT04549142
Title: Immune Tolerance Dysfunction in Pregnancy Due to Ambient Air Pollution
Brief Title: Immune Tolerance Dysfunction in Pregnancy Due to Ambient Air Pollution Exposure
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH); Duke University (Other)
Responsible Party: Principal Investigator, R. Sharon Chinthrajah, Associate Professor of Medicine, Stanford University
Other Study IDs: IRB-56622; R01ES032253 (NIH)
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Air Pollution; Pregnancy
Keywords: immune function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pregnant women- high level pollution: Exposed to high levels of pollution (PM2.5)
  Interventions: Other: There is no intervention
- Pregnant women- low level pollution: Exposed to low levels of pollution (PM2.5)
  Interventions: Other: There is no intervention
- Non-pregnant women-high level pollution: Exposed to high levels of pollution (PM2.5)
  Interventions: Other: There is no intervention
- Non-pregnant women-low level pollution: exposed to low levels of pollution (PM2.5)
  Interventions: Other: There is no intervention

INTERVENTIONS:
Other: There is no intervention — There is no intervention

SUMMARY:
The purpose of this project is to study the effects of air pollution toxicants on pregnant mothers' immune health during and after pregnancy.

Using already collected samples, this study proposes to evaluate changes in immune function in response to air pollution with the use of innovative technologies, to identify the drivers of immune dysfunction and potential modifiable factors, and to determine how these immune findings are associated with pollution exposure and outcomes of disease.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women: at 18-25 weeks gestation at time of eligibility screening and baseline visit

Exclusion Criteria:

* Having smoked more than 50 cigarettes during pregnancy
* A history of autoimmune diseases, HIV or cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women at 18-25 weeks gestation and non-pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Difference in immune cell subset identity and function in pregnant vs. non pregnant women exposed to high vs. low pollution over time | 3 years
Identify the epigenetic molecular mechanisms driving immune dysfunction in pregnancy vs. no pregnancy with high vs. low PM2.5 exposure over time | 3 years
Map T cell receptor diversity to immune dysfunction in pregnancy vs non pregnancy with high vs. low PM2.5 exposure over time | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: R. Sharon Chinthrajah, MD, Principal Investigator — Stanford, Sean N Parker Center for Allergy and Asthma Center at Stanford
Locations (1):
- Sean N. Parker Center for Allergy & Asthma Research at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No